CLINICAL TRIAL: NCT01286948
Title: A Randomized, Cross-over, Clinical Trial to Assess the Prevention of Ovulation Achieved by Single Intra-vaginal Administration of 0.75 mg Levonorgestrel (LNG) Gel (Levogel) as Compared to 1.5 mg Oral LNG
Brief Title: Prevention of Ovulation Achieved by Single Intra-vaginal Administration of Levogel as Compared to Oral LNG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol # 441
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Female Contraception
Keywords: LNG gel; oral LNG; follicle rupture; intra-vaginal administration; growth of the leading follicle; preovulatory peak of serum luteinizing hormone; characteristics of the cervical mucus; serum levels of estradiol (E2) and progesterone (P)
MeSH Terms: interventions — Levonorgestrel; Gels

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levonorgestrel (LNG) gel (Levogel) (Active Comparator): This is a randomized study with a cross-over design comparing two single dose treatment sequences of either Levogel (LNG vaginal gel 0.750 mg/4g) or oral LNG (1.5mg).
  All women with a leading follicle diameter of ≥18 mm will be randomized to treatment with a single intra-vaginal application of LNG gel or oral LNG. After a washout cycle, the women will be crossed over to receive the other treatment and the study procedures will be repeated.
  Interventions: Drug: Levonorgestrel (LNG) gel (Levogel) and oral LNG (Plan B)
- oral LNG (1.5mg) (Active Comparator): This is a randomized study with a cross-over design comparing two single dose treatment sequences of either Levogel (LNG vaginal gel 0.750 mg/4g) or oral LNG (1.5mg).
  All women with a leading follicle diameter of ≥18 mm will be randomized to treatment with a single intra-vaginal application of LNG gel or oral LNG. After a washout cycle, the women will be crossed over to receive the other treatment and the study procedures will be repeated.
  Interventions: Drug: Levonorgestrel (LNG) gel (Levogel) and oral LNG (Plan B)

INTERVENTIONS:
Drug: Levonorgestrel (LNG) gel (Levogel) and oral LNG (Plan B) — This is a randomized study with a cross-over design comparing two single dose treatment sequences of either Levogel (LNG vaginal gel 0.750 mg/4g) or oral LNG (1.5mg).
  All women with a leading follicle diameter of ≥18 mm will be randomized to treatment with a single intra-vaginal application of LNG gel or oral LNG. After a washout cycle, the women will be crossed over to receive the other treatment and the study procedures will be repeated.

SUMMARY:
It has been proposed that levonorgestrel (LNG) in a vaginal gel could be used as an 'on demand' contraceptive when used before coitus. Levonorgestrel was selected as it is a component of many approved oral contraceptive pills and also it is the active agent in Plan B, an FDA-approved regimen for emergency contraception (EC). In previous studies it was demonstrated that an LNG vaginal gel was absorbed and was effective in preventing follicular rupture. The overall proportion of cycles with lack of follicular rupture within 5 days of LNG administration or with ovulatory dysfunction (follicle rupture preceded by an inadequate LH surge) was 96% for LNG gel and 39% in the inert gel cycles (control group).

DETAILED DESCRIPTION:
A dose of 0.75mg of LNG in a vaginal gel was shown to prevent ovulation in a higher percentage than what has been observed with oral LNG at the approved doses for EC of 1.5mg. Results from a study with a1.5 mg LNG oral dose or a single 0 ,75mg dose demonstrated that the proportion of cycles without follicle rupture or ovulatory dysfunction within 5 days was 86% and 79% respectively (Croxatto et al, 2004) , whereas lack of follicular rupture or the presencr of ovulatory dsyfunction was 96% with administration of a LNG gel formulation. In the group of women with follicle size ≥18mm the gel induced 50% ovulation suppression while oral LNG in previous studies blocked only 16% of ovulation in the same follicle size group . These encouraging results could be explained by higher bioavailability of LNG when administered vaginally. This comparison was made using historical data from another study; therefore this study will compare vaginal administration of LNG to oral in a direct cross-over comparative study.

LNG is known to affect the cervical mucus by making it hostile to sperm penetration and its effect may appear after only a few hours following oral administration (Kesseru, 1984; Brache, unpublished observations). Application of LNG gel in the vagina close to the cervical os may exert a direct effect on the cervical mucus. The potential local action of LNG on the cervical mucus may be another important mechanism by which protection is conferred to women who do not experience ovulation suppression.

An "on demand" precoital contraceptive is an attractive alternative to the post-coital emergency contraception currently available, especially due to the higher efficacy of this route of administration on ovulation suppression as compared with oral tablets of LNG. Should the present study confirm the superiority of vaginal administration of half the dose of the oral dose of LNG approved for emergency contraception, further development of that formulation and method would be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 21-39 years with regular menstrual cycles (25-35 days) and not at risk of pregnancy.

Exclusion Criteria:

* All contraindications to the use of progestins

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Comparison of LNG gel and oral LNG on follicle rupture | 1 year
  The main objective of the study is to compare the effect of LNG gel and oral LNG on follicle rupture as assessed by ultrasound.

SECONDARY OUTCOMES:
Evaluate effect of single intra-vaginal administration | 1 year
  The secondary objectives are to evaluate the effect of single intra-vaginal administration of LNG gel or oral LNG on the:
  * growth of the leading follicle
  * suppression of the preovulatory peak of serum luteinizing hormone (LH)
  * characteristics of the cervical mucus
  * serum levels of estradiol (E2) and progesterone (P)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Brache, Lic., Principal Investigator — Profamilia; Regine Sitruk-Ware, PhD., Principal Investigator — Population Council; María José Miranda Gaete, MD, Principal Investigator — Instituto Chileno de Medicina Reproductiva
Locations (2):
- Instituto Chileno de Medicina Reproductiva, José Victorino Lastarria 29, Santiago Metropolitan, Chile
- Profamilia, Socorro Sanchez No. 160, Santo Domingo Province, Dominican Republic